CLINICAL TRIAL: NCT06299930
Title: Locoregional Recurrence After Neoadjuvant Versus Adjuvant Chemotherapy Based on Tumor Subtypes in Patients With Early-stage Breast Cancer: A Multi-institutional Retrospective Cohort Study
Brief Title: Locoregional Recurrence After Neoadjuvant Versus Adjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonshik Han, Clinical Professor, Seoul National University Hospital
Other Study IDs: LRR after NACT vs ACT
Record Dates: First submitted 2024-02-14; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemotherapy (NACT) group: Patients who administered chemotherapy before surgery
  Interventions: Procedure: Neoadjuvant chemotherapy
- Adjuvant chemotherapy (ACT) group: Patients who administered chemotherapy after surgery
  Interventions: Procedure: Adjuvant chemotherapy

INTERVENTIONS:
Procedure: Neoadjuvant chemotherapy — Patients received neoadjuvant chemotherapy (either taxane-or anthracycline-based, or any cytotoxic chemotherapy) , followed by surgery and radiotherapy
  Other Names: NACT
  Groups: Neoadjuvant chemotherapy (NACT) group
Procedure: Adjuvant chemotherapy — Patients received adjuvant chemotherapy (either taxane-or anthracycline-based, or any cytotoxic chemotherapy) after surgery, followed by radiotherapy
  Other Names: ACT
  Groups: Adjuvant chemotherapy (ACT) group

SUMMARY:
Neoadjuvant chemotherapy (NACT) for early-stage breast cancer is associated with an increased risk of locoregional recurrence (LRR). However, few studies have conducted subgroup analyses of patients with various molecular subtypes, which are one of the determinant factors for treatments. The aim of the study is to investigate whether the risk of LRR after NACT varies across tumor subtypes. The investigators retrospectively reviewed the medical records of female breast cancer patients who underwent breast-conserving surgery at three institutions between January 1, 2004, and Dec 31, 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent breast-conserving surgery for invasive breast cancer between 2004 and 2018

Exclusion Criteria:

* Total mastectomy
* No pre- or postoperative chemotherapy
* No radiation therapy
* Bilateral breast cancer
* Male breast cancer patients
* Secondary breast cancer
* Metachronous or synchronous cancers

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients who underwent breast-conserving surgery for breast cancer between January 1, 2004 and December 31, 2018 at the three leading hospitals in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 10328 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Locoregional recurrence-free survival (LRR) | Defined as the time interval between the date of initial administration of chemotherapy and date of pathological or radiological confirmation of LRR, assessed up to 120 months
  Time interval between the date of initial administration of chemotherapy and date of pathological or radiological confirmation of locoregional recurrence

SECONDARY OUTCOMES:
Distant metastasis-free survival | Defined as the time interval between the date of initial administration of chemotherapy and date of pathological or radiological confirmation of distant metastasis, assessed up to 120 months
  Time interval between the date of initial administration of chemotherapy and date of pathological or radiological confirmation of distant metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT06299930/Prot_SAP_000.pdf